CLINICAL TRIAL: NCT04176640
Title: Quantifying Brain Injury on Computed Tomography in Hospitalized Children: a Prospective Trial
Brief Title: Quantifying Brain Injury on Computed Tomography in Hospitalized Children
Acronym: QBIct
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Anne-Marie Guerguerian, Senior Scientist, The Hospital for Sick Children
Other Study IDs: REB1000050054
Record Dates: First submitted 2019-10-24; First posted 2019-11-25 (Actual); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Trauma, Brain; Pediatric
Keywords: pediatric traumatic brain injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Lay Summary:

To evaluate a novel early diagnostic tool for hospitalized children with traumatic brain injury.

The Problem: Children who present with decreased level of consciousness after injury require urgent medical attention determined by the type and the severity of injury. Unfortunately, history and physical findings are often unreliable in the first hours after hospitalization, the period in which urgent management decisions must be made for their treatment.

The Solution: A promising tool developed for measuring detectable evidence of traumatic brain injury on routine brain scans. The tool combines features invisible to the human eye but detectable by computer software with expert knowledge.This study will evaluate how well the tool can perform in a real health care setting. It is believed that it will greatly improve the efficacy and quality of care provided to children after traumatic brain injury.

DETAILED DESCRIPTION:
To evaluate a novel early neuroimaging diagnostic tool for hospitalized children with traumatic brain injury.

This tool is used to detect evidence of traumatic brain injury on routine brain scans. The tool combines features invisible to the human eye but detectable by computer software with expert knowledge.This study will evaluate how well the tool can perform in a real health care setting. It is believed that it will greatly improve the efficacy and quality of care provided to children after traumatic brain injury.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized with TBI
* Age: less than 18 years of age who undergoes routine head CT in the acute period with any severity of injury based on Glasgow Coma Scale score (3 to15).

Exclusion Criteria:

* Non hospitalized
* Non traumatic brain injury

Ages: 1 Day to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Hospitalized children with traumatic brain injury
Sampling Method: Non-Probability Sample
Enrollment: 425 (Actual)
Dates: Start 2015-10-20 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
To measure if QBIct predicts the development of new cerebral dysfunction measured on the Glasgow Outcome Scale Extended for Pediatrics score | 30 days
  GOSE for Pediatrics score is the reference standard for measuring traumatic brain injury (TBI) outcome. GOSE-P is a NINDS Common Data Element for functional outcome that rates patient status into one of eight categories: Dead, Vegetative State, Lower severe disability, Upper severe Disability, Lower moderate disability, Upper moderate Disability, Lower good recovery or Upper good Recovery. Minimum score = 1, Maximum score = 8
  Level 1 = Dead Level 2 = Vegetative State Level 3 = Low Severe Disability Level 4 = Upper Severe Disability Level 5 = Lower Moderate Disability Level 6 = Upper Moderate Disability Level 7 = Low Good Recovery Level 8 = Upper Good Recovery

SECONDARY OUTCOMES:
To determine if QBIct tool predicts secondary clinical outcomes | 90 days
  Clinical outcomes were defined as intracranial hypertension and/or, need for neurosurgical intervention and/or early mortality.
To determine if QBIct tool predicts recovery endpoints. | 90 days
  Endpoints were defined by global functional outcomes, mechanical ventilation days, and intensive care days, hospital days and/or home from school days.
  Global functional outcomes will be measured using Vineland-II. Vineland-II is a standardized psychological tool used to measure 4 major aspects of adaptive functioning: Communication, Daily Living Skills, Socialization and Motor Skills. It measures the personal and social skills of individuals from birth through adulthood. Because adaptive behavior refers to an individual's typical performance of the day-to-day activities required for personal and social sufficiency, these scales assess what a person actually does, rather than what he or she is able to do.
  In order to determine the level of an individual's adaptive behavior, someone who is familiar with that individual, such as a parent or caregiver, is asked to describe his activities. Those activities are then compared to those of ot

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Marie Guerguerian, Principal Investigator — The Hospital for Sick Children, University of Toronto

REFERENCES:
- See also: QBI CT Web Site — https://lab.research.sickkids.ca/qbict/